CLINICAL TRIAL: NCT06846905
Title: Cost-utility Analysis of Ambulatory Dose Escalation of Bispecific Antibodies in Multiple Myeloma.
Acronym: AmbuSpé
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0480
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Multiple myeloma; Neoplasms; Plasma Cell; Antineoplastic Agents; Antibodies Bispecific; Outpatient Care
MeSH Terms: conditions — Multiple Myeloma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Outpatient step-up dose procedure: Patients treated on an outpatient procedure if it's clinically feasible (good condition general, no rapid progression or major tumor burden, no current infection) and logistics (lived within 30 minutes from the IUCT Oncopole for 48 hours after each step-up dose)
- Conventional procedure: Patients who do not meet the conditions for outpatient care and justify hospitalization in a conventional unit for dose escalation

SUMMARY:
Multiple myeloma is the second most common haematological cancer. Recent innovations have made it possible for relapsed/refractory patients to benefit from the innovative immunotherapy of bispecific antibodies. These antibodies stimulate the immune system to attack tumour cells. The treatment involves an escalating dose of three subcutaneous injections every 2 to 4 days for a total of about 10 days, followed by a weekly treatment phase.

The University Hospital of Toulouse was the first centre in France to offer outpatient dose escalation for this innovative treatment. This form of treatment depends on clinical and logistical feasibility. Where appropriate, patients are treated in a conventional unit. An analysis carried out at Toulouse University Hospital suggests a response to treatment, with no increased risk of complications in the outpatient setting. Patients' quality of life may also be unaffected. In addition, given the increasing demand for care in a context of finite resources, the economic evaluation of healthcare initiatives is becoming essential if we are to maintain a high-quality healthcare system that is accessible to all.

DETAILED DESCRIPTION:
The study has two arms: patients treated in the outpatient unit and patients treated in the conventional unit. The prospective data collection is based on quality of life at three time points during the dose escalation phase. The following questionnaires will be used: EQ-5D-5L for utility analysis, QLQ-C30 validated in cancer patients and QLQ MY20 validated in multiple myeloma patients. Clinical data will be collected as well as economic data related to hospital stays.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed and/or refractory multiple myeloma
* Treated with teclistamab, elranatamab ou talquetamab
* More than 18 years old
* Having received the information from the study and not having objected to participate
* Day hospital care in case of clinical feasibility (good general condition, no rapid progression or major tumor burden, no current infection) and logistics (accommodated less than 30 minutes from the IUCT Oncopole for 48 hours after each dose escalation) or in conventional hospitalization at the IUCT Oncopole

Exclusion Criteria:

* Illiterate subjects or those with a language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study proposed during haematology consultation at the IUCT-Oncopole, detailing the care plan.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficiency | 30 days
  Cost of the procedure for health system and quality-adjusted life year calculated from the generic EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Toulouse, Toulouse, France